CLINICAL TRIAL: NCT02252250
Title: A Prospective Cohort Study of Transanal Laparoscopic Total Mesentery Excision Versus Conventional Laparoscopic Surgery for Rectal Cancer
Brief Title: Transanal Total Mesorectal Excision Versus Laparoscopic TME for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Weidong Tong, Dr, Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20141056
Record Dates: First submitted 2014-09-23; First posted 2014-09-30 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Rectal Neoplasms
Keywords: rectal cancer; laparoscopic; taTME; TME
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional laparoscopic (Active Comparator): conventional laparoscopic total mesentery excision surgery for rectal cancer.
  Interventions: Procedure: conventional laparoscopic total mesentery excision
- Transanal hybrid-laparoscopic (Experimental): Transanal hybrid-laparoscopic total mesentery excision surgery for rectal cancer.
  Interventions: Procedure: transanal hybrid-laparoscopic total mesentery excision

INTERVENTIONS:
Procedure: conventional laparoscopic total mesentery excision — conventional laparoscopic total mesentery excision
  Other Names: LTME
  Arms: conventional laparoscopic
Procedure: transanal hybrid-laparoscopic total mesentery excision — transanal laparoscopic total mesentery excision for rectal cancer. Mobilize the rectum from down- to-up. Then, set a single incision laparoscopic surgery (SILS) port at the right-low abdomen to resect the lymph nodes of IMA.
  Other Names: TLTME
  Arms: Transanal hybrid-laparoscopic

SUMMARY:
To investigates the feasibility, practicability, safety and subjective as well as functional outcome of transanal minimal invasive surgery toal mesentery excision for rectal cancer.

DETAILED DESCRIPTION:
Natural orifice transluminal endoscopic surgery (NOTES) give the opportunity to reduce surgical access trauma leading to a more painless surgery and enhancing a fast postoperative recovery. Experience with transanal minimal invasive surgery(TAMIS) for rectal cancer show that such NOTES procedures are feasible and safe. And also, lots of experimental studies and small case series reporting the feasibility of transanal anterior resection with single incision laparoscopic surgery(SILS) port or other devices. However any prospective feasibility study demonstrating the safety of the procedure and functional outcomes (sphincter function, sexual function, QOF) are missing. This study investigates the feasibility, practicability, safety and subjective as well as functional outcome of transanal minimal invasive total mesentery excision for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven adenocarcinoma of the rectum
* Eligible to undergo conventional laparoscopic low anterior resection or transanal hybrid-laparoscopic low anterior resection with or without a temporary diverting stoma
* Node negative (N0), T1 (high risk features), T2 and T3 rectal cancer on pelvic MRI
* Closest distance between tumor edge and mesorectal fascia 5mm or more based on pelvic MRI
* Rectal cancer located 3-10 cm from the anal verge

Exclusion Criteria:

* Metastasis
* Obstructing rectal cancer
* Synchronous colon cancer
* T4 rectal cancer not treated preoperatively with full-course chemoradiation
* Pregnant or breast-feeding
* Receiving any other study agents
* Fecal incontinence
* History of prior colorectal cancer
* History of inflammatory bowel disease
* History of pelvic radiation
* BMI > 40
* Large uterine fibroids
* Uncontrolled intercurrent illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Adequacy of the total mesorectal excision(TME) based on standard guidelines on pathologic evaluation of TME specimens. | 1-6 years
  Lymph nodes number; rate of positive circumferential resection margin(CRM);

SECONDARY OUTCOMES:
Incidence of 30-day perioperative complications including intraoperative, and postoperative complications | 0-30 days
  bleeding, injury of adjacent organs, ileus, leakage, infection
Incidence of long-term complications | 1-6 years
  incision hernia,
Oncologic outcomes in subjects receiving transanal hybrid-laparoscopic total mesentery excision. | 1-6 years
  overall survive rate and disease free survive rate of 3 and 5 years; recurrence rate

OTHER OUTCOMES:
defecating functional outcomes | 1-6 years
  constipation score and incontinence score
sexual functional outcomes | 1-6 years
  We examine before operation, 3 months after, 6 months after, 12 months after, 24 months after operation, by questionnaires (International Index of Erectile Function (IIEF)
Quality of life outcomes evaluation | 1-6 years
  We examine before operation, 3 months after, 6 months after, 12 months after, 24 months after operation, by questionnaires (Short Form-36 (SF36) and Gastro-Intestinal Functional Outcome(GIFO)) .

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Tong, Prof, Principal Investigator — Daping Hospital, Third Military Medical University
Locations (1):
- Daping hospital, Chongqing, Chongqing Municipality, China